CLINICAL TRIAL: NCT05752188
Title: Prognostic Value of Cardiovascular Risk of Soluble Suppression of Tumorigenesis-2 and High Sensitivity Troponin I in Patients With Acute Chest Pain
Brief Title: Prognostic Value of Cardiovascular Risk of sST2 and Troponin I-hs in Patients With Acute Chest Pain
Acronym: sST2
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Baroni Silvia, Confirmed researcher - Adjunct Professor-M.D., Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3477
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Acute Chest Pain; Acute Coronary Syndrome
Keywords: Troponin; sST2
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — residual serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Multimarker approach in acute coronary syndrome — The main objective of the study is to evaluate the prognostic role of the biochemical marker sST2 in patients attending the Emergency Department of our hospital with acute chest pain with suspected acute coronary syndrome.

SUMMARY:
The role of the sST2 biomarker has been widely explored in heart failure, so much so that it was included in the AHA guidelines in 2013 and 2017. Recently, several studies are proposing a role of sST2 in the prognostic stratification of patients with Acute Coronary Syndrome and ischemic heart disease, in association with other biomarkers even proposing a possible therapeutic differentiation. The combined use of sST2 with high-sensitivity troponins could be a promising strategy to identify those patients who, despite having early rule-out after evaluation at the Emergency Department, have a higher risk of onset of cardiovascular events in the medium-long term.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Chest pain of presumable cardiac origin and uncertain etiological diagnosis
* ECG not diagnostic for ischemia
* troponin values within normal ranges

Exclusion Criteria:

* STEMI myocardial infarction
* Sepsis and viral infections
* Patients with ECG abnormalities that make it uninterpretable for ischemic purposes
* Patients with previous coronary events
* History of heart failure
* Known diagnosis of cardiovascular disease, acute or chronic, including pericarditis, myocarditis
* Conditions involving sST2 elevations unrelated to cardiac causes, particularly acute/chronic inflammatory or fibrotic conditions (inflammatory bowel disease, malignancy, moderate to severe pulmonary fibrosis, chronic liver disease; autoimmune disorders)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The evaluation of the efficacy of the sST2 and cTNI HS biomarkers will be evaluated retrospectively without altering the normal diagnostic and therapeutic procedure in the recruited patients.
  The results of sST2 and Troponins will then be evaluated on the basis of the clinical outcomes obtained by telephone interview with the patient carried out at 1 year.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-07-03 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Evaluate sST2 predictive value's | 24 months
  Evaluate the medium-long term (1 year) predictive value of the sST2 biomarker in the heart patients attending at the Emergency Department for non-STEMI Acute Chest Pain.

SECONDARY OUTCOMES:
Compare sST2 prognostic value with troponins | 24 months
  Compare the prognostic value of the new biomarker with highly sensitive troponins, for which there is already evidence in the literature
Create a multiparametric algorithm/score | 36 months
  Integrate the sST2 values in a multiparametric algorithm/score for the differential diagnosis and risk stratification in medium/long-term complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Silvia Baroni, Roma, Italy

REFERENCES:
- [Background] Aimo A, Vergaro G, Ripoli A, Bayes-Genis A, Pascual Figal DA, de Boer RA, Lassus J, Mebazaa A, Gayat E, Breidthardt T, Sabti Z, Mueller C, Brunner-La Rocca HP, Tang WH, Grodin JL, Zhang Y, Bettencourt P, Maisel AS, Passino C, Januzzi JL, Emdin M. Meta-Analysis of Soluble Suppression of Tumorigenicity-2 and Prognosis in Acute Heart Failure. JACC Heart Fail. 2017 Apr;5(4):287-296. doi: 10.1016/j.jchf.2016.12.016. Epub 2017 Feb 8. PMID 28189578
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). Circulation. 2018 Nov 13;138(20):e618-e651. doi: 10.1161/CIR.0000000000000617. No abstract available. PMID 30571511
- [Background] Roffi M, Patrono C, Collet JP, Mueller C, Valgimigli M, Andreotti F, Bax JJ, Borger MA, Brotons C, Chew DP, Gencer B, Hasenfuss G, Kjeldsen K, Lancellotti P, Landmesser U, Mehilli J, Mukherjee D, Storey RF, Windecker S; ESC Scientific Document Group. 2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: Task Force for the Management of Acute Coronary Syndromes in Patients Presenting without Persistent ST-Segment Elevation of the European Society of Cardiology (ESC). Eur Heart J. 2016 Jan 14;37(3):267-315. doi: 10.1093/eurheartj/ehv320. Epub 2015 Aug 29. No abstract available. PMID 26320110
- [Background] Reichlin T, Schindler C, Drexler B, Twerenbold R, Reiter M, Zellweger C, Moehring B, Ziller R, Hoeller R, Rubini Gimenez M, Haaf P, Potocki M, Wildi K, Balmelli C, Freese M, Stelzig C, Freidank H, Osswald S, Mueller C. One-hour rule-out and rule-in of acute myocardial infarction using high-sensitivity cardiac troponin T. Arch Intern Med. 2012 Sep 10;172(16):1211-8. doi: 10.1001/archinternmed.2012.3698. PMID 22892889
- [Background] Januzzi JL, Pascual-Figal D, Daniels LB. ST2 testing for chronic heart failure therapy monitoring: the International ST2 Consensus Panel. Am J Cardiol. 2015 Apr 2;115(7 Suppl):70B-5B. doi: 10.1016/j.amjcard.2015.01.044. Epub 2015 Jan 24. PMID 25670638
- [Background] Sabatine MS, Morrow DA, Higgins LJ, MacGillivray C, Guo W, Bode C, Rifai N, Cannon CP, Gerszten RE, Lee RT. Complementary roles for biomarkers of biomechanical strain ST2 and N-terminal prohormone B-type natriuretic peptide in patients with ST-elevation myocardial infarction. Circulation. 2008 Apr 15;117(15):1936-44. doi: 10.1161/CIRCULATIONAHA.107.728022. Epub 2008 Mar 31. PMID 18378613